CLINICAL TRIAL: NCT01679847
Title: Blood Brain Barrier Penetration and Pharmacokinetics of the Elemene in Malignant Patients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dalian Holley Kingkong Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: HSZL201001
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Cancer
Keywords: Elemene; pharmacokinetics; Blood-brain barrier
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples Without DNA — Plasma and Cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to elucidate the pharmacokinetics and the blood-brain barrier penetration of the elemene.

ELIGIBILITY:
Inclusion Criteria:

* histopathological or cytopathology diagnosis of malignancy
* heart, liver and renal function is normal
* Expected survival time is more than 3 months
* Signed informed consent

exclusion Criteria:

* non cancer patient
* accepted elemene administration in 1 month
* Expected survival time is less than 3 months
* no Signed informed consent
* heart, liver and renal function is abnormal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: malignant patients
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-04 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
blood and cerebrospinal fluid concentration | 0，0.25，0.5，1，1.5，2，3，3.5，4，6，8，12 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: liang xiaohua, phD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality, China